CLINICAL TRIAL: NCT03697148
Title: Multiparametric MRI (mpMRI) for Preoperative Staging and Treatment Planning for Newly-Diagnosed Prostate Cancer
Brief Title: Multiparametric MRI in Evaluating Cancer Stage and Helping Treatment Planning in Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EA8171; NCI-2017-01997 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8171 (Other: ECOG-ACRIN Cancer Research Group); EA8171 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2018-07-10; First posted 2018-10-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Diagnostic (mpMRI) (Experimental): Patients undergo mpMRI within 3 months prior to schedule surgery.
  Interventions: Diagnostic Test: Multiparametric Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Multiparametric Magnetic Resonance Imaging — Undergo mpMRI
  Other Names: MP-MRI; Multi-parametric MRI; Multiparametric MRI

SUMMARY:
This phase II trial studies how well multiparametric magnetic resonance imaging (MRI) works in evaluating cancer stage and helping treatment planning in patients with prostate cancer. Multiparametric MRI may be useful for evaluating the type of cancer in finding aggressive disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the diagnostic performance as quantified by the area under the ROC curve to detect aggressive prostate cancer.

II. To develop a risk prediction model by incorporating overall PI-RADS, PSA, Gleason score and clinical stage to predict the presence of aggressive prostate cancer.

SECONDARY OBJECTIVES:

I. To evaluate the diagnostic performance of the individual PI-RADS score of each MRI parameter (T2W, DWI and DCE), as determined by local imaging review.

TERTIARY OBJECTIVES:

I. All clinical data including magnetic resonance (MR) images will be banked for future exploratory research aims.

OUTLINE:

Patients undergo mpMRI within 3 months prior to schedule surgery.

After completion of study, patients are followed up until radical prostatectomy pathology is reported and finalized.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed with prostate cancer for whom definitive surgical treatment is indicated

Exclusion Criteria:

* Not suitable to undergo MRI or receive gadolinium-based contrast agent (severe, untreatable claustrophobia; MRI-incompatible metallic objects or implanted medical devices; renal failure; weight greater than allowable by scanner per institutional standard practice)
* Prior surgical and/or non-surgical treatment for prostate cancer
* Prior hip replacement or other major pelvic surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of overall prostate imaging reporting and data system (PI-RADS) score | Up to 2 years
  Will estimate the diagnostic performance as quantified by the area under the ROC curve.
Risk prediction model | Up to 2 years
  To estimate the predictive performance of a model for predicting clinically significant prostate cancer on the basis of the overall PI-RADS, PSA, Gleason score and clinical stage.

SECONDARY OUTCOMES:
Diagnostic performance of the individual prostate imaging reporting and data system (PI-RADS) score | Up to 2 years
  Will estimate the diagnostic performance as quantified by the area under the ROC curve.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Tempany-Afdhal, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (44):
- United States (44):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Yale University, New Haven, Connecticut
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Straub Pearlridge Clinic, ‘Aiea, Hawaii
  - Midwestern Regional Medical Center, Zion, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin